CLINICAL TRIAL: NCT06183892
Title: Prospective, Multicenter Clinical Study of Prolonged-release Tacrolimus in Stable Pediatric Liver Transplant Recipients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Renji-LY2023-076-B
Record Dates: First submitted 2023-06-22; First posted 2023-12-28 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Liver Transplant
Keywords: liver transplant; pediatric liver transplant; tacrolimus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prolonged-release tacrolimus (Experimental)
  Interventions: Drug: Tacrolimus Sustained-release Capsules

INTERVENTIONS:
Drug: Tacrolimus Sustained-release Capsules — Immediate-release tacrolimus for at least 3 months after liver transplantation, and then convert to tacrolimus sustained-release capsules at a ratio of 1:1 to 1:1.2; Take the medicine once a day on an empty stomach in the morning.
  (The specific medication plan is decided by the clinician according to the actual situation)

SUMMARY:
This study aims to explore the effects of tacrolimus sustained-release capsules on the incidence of biopsy-proven acute rejection(BPAR) and fibrosis in pediatric liver transplant recipients.

DETAILED DESCRIPTION:
Tacrolimus is a commonly used immunosuppressant after liver transplantation. However, with increased postoperative time and a decline in postoperative compliance, some children may miss medication, leading to acute rejection. Repeated rejection can cause fibrosis of the transplanted liver, seriously impacting graft function and even postoperative survival, sometimes resulting in the need for a second liver transplant. In adult liver transplant recipients, tacrolimus sustained-release capsules have been shown to significantly improve overall and transplanted liver survival compared to conventional formulations (immediate-release tacrolimus，taken twice daily). Therefore, this study aims to explore the effects of tacrolimus sustained-release capsules on the incidence of biopsy-proven acute rejection(BPAR) and fibrosis in pediatric liver transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

1. Children (≤18 years old) who have undergone liver transplantation, with no gender limitations;
2. Able to completely swallow capsules;
3. Have been using immediate-release tacrolimus for at least three months prior to study enrollment;
4. Have normal blood count, liver and kidney function, coagulation function, and considered clinically stable by researchers;
5. Undergo a programmed liver biopsy;

Exclusion Criteria:

1. Multi-organ combined transplantation or multiple liver transplantation;
2. Adjuvant liver transplantation or use of bioartificial liver therapy;
3. ABO incompatible children with liver transplantation;
4. Allergic to tacrolimus;
5. Participation in any other clinical study within 3 months prior to enrollment;
6. Use of tacrolimus sustained release capsules before enrollment;
7. Tacrolimus trough concentration lower than 3.5 ng/ml at the time of screening;

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of biopsy-confirmed acute rejection (BPAR) | 12 months
  biopsy-confirmed acute rejection (BPAR) would be evaluated by the international Banff classification
Incidence of allograft liver fibrosis | 12 months
  allograft liver fibrosis would be evaluated by LAFSc

SECONDARY OUTCOMES:
Liver function | 12 months
  alanine transaminase (ALT) and aspartate transaminase (AST), serum bilirubin, prothrombin time (PT), and albumin within and 12 months after conversion
Kidney function | 12 months
  creatinine (Cr) and BUN within and 12 months after conversion
Liver allograft survival rate | 12 months
  Liver allograft survival rate at 12 months after conversion
The rate of drug change | 12 months
  The rate of drug change caused by ultrasonic diagnosis and abnormal liver function index suspected AR (from tacrolimus sustained release to other CNI drugs)
Incidence of infection | 12 months
  Incidence of infection (viral, bacterial and fungal) at 12 months after conversion

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Xia, Prof. MD, Study Chair — Dept. Liver Surgery, Renji Hospital, School of Medicine, SJTU; Hao Feng, MD., Ph.D, Principal Investigator — Dept. Liver Surgery, Renji Hospital, School of Medicine, SJTU
Locations (1):
- Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No